CLINICAL TRIAL: NCT04376398
Title: Survey on Patients With Suspected or Confirmed COVID-19 Requiring Anesthesia Care for Their Intervention
Brief Title: Survey: COVID-19 Patients Managed in the Operating Theatre of Belgian Hospitals
Acronym: COVID
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Society for Anesthesia and Resuscitation of Belgium (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVID-ANESTHESIO
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Any pediatric or adult patient with COVID-19 or suspected of COVID-19 scheduled for any intervention

SUMMARY:
COVID-19 pandemic has an important impact on the health care provided by the anesthesiologists. Different societies of anesthesiology have provided guidelines and recommendations on how to manage patients who have been tested positive for COVID-19 or suspected to be infected. It is therefore important to know whether these guidelines have been implemented or were possible to be implemented. Otherwise patients who are presenting COVID-19 often show pulmonary complications. The airway management and the ventilation management of these patients can be therefore challenging and can possibly influence their outcome. It is thus important to obtain a large database with information about the characteristics of these patients, how these patients have been managed and their in-hospital outcome. Information regarding the correct implementation of guidelines is as well necessary for future guidance of health care providers.

ELIGIBILITY:
Inclusion Criteria:

* All patients (pediatric/adults/parturients) who are tested positive for COVID-19 or who are suspected to be infected

Exclusion Criteria: No oral consent

-

Ages: 1 Hour to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pediatric and adult patients who are tested positive for COVID-19 or who are suspected to be infected and who require anesthesia care for their intervention
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Global evaluation of the implication of the Belgian anesthesiologists during COVID-19 pandemic | 30 days
  To evaluate whether Belgian anesthesiologists have followed or could follow the recommendations regarding the management of COVID-19 patients and what were the characteristics of these patients and how they have been managed and what were their outcomes

SECONDARY OUTCOMES:
If any compare our results with other countries | 4 weeks
  To compare the descriptives and the outcome data of our patients with other countries

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
All data will be provided to the Society for Anesthesia and Resuscitation of Belgium